CLINICAL TRIAL: NCT00934271
Title: Fractionated Stereotactic Radiotherapy in Patients With Acromegaly. Single Centre Experience
Brief Title: Fractionated Stereotactic Radiotherapy in Patients With Acromegaly
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, chief Physician, Rigshospitalet, Denmark
Other Study IDs: FSRT-SR-UFR
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Acromegaly
Keywords: acromegaly; irradiation; remission; pituitary function
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fractionated stereotactic radiotherapy: patients with active acromegaly
  Interventions: Radiation: fractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: fractionated stereotactic radiotherapy — Audit of outcome

SUMMARY:
Hypothesis: Fractionated stereotactic radiotherapy is a safe therapy for treatment of patients with acromegaly in terms of both tumour control and biochemical remission

DETAILED DESCRIPTION:
An audit was done on 34 patients with acromegaly (consecutive cohorte) treated with fractionated stereotactic radiotherapy in Rigshospitalet/National University Hospital, Copenhagen, Denmark. All patients had MR control regularly to monitor tunour control, and biochemical control assessed by growth hormone measurements during an oral glucose tolerance test. Furthermore all other pituitary axes were tested for sufficiency and concomitant medication likewise registered. The 7 year interim analysis demonstrated an acceptable tumour control and biochemical remission profile, and most patient had subsequent withdrawal of somatostatin analogue- and growth hormone receptor antagonis therapy. The observational study will continue with a new update in approx 2 years

ELIGIBILITY:
Inclusion Criteria:

adults active acromegaly pituitary tumour on MRI biochemical activity -

Exclusion Criteria:

pregnancy no visible tumour on MRI

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 34 patients with active acromegaly despite medical therapy
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2002-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Tumour control by pituitary MRI | 7 years

SECONDARY OUTCOMES:
biochemical remission | 10 years
Affection of other pituitary axes | 10 years
withdrawal of somatostatin analogue and growth hormone receptor antagomist | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Department of Medical Endocrinology, Copenhagen, Denmark